CLINICAL TRIAL: NCT04112511
Title: Study of Myocardial Deformation Parameters in Patients With Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Zegkos, Medical Doctor, Resident in Cardiology, AHEPA University Hospital
Other Study IDs: 4045PHD
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate the potential correlations of global longitudinal strain and peak left atrial strain, measured by speckle tracking echocardiography with the severity of hypertrophic cardiomyopathy and the risk for arrhythmias.

Specifically the investigational questions are:

1. Is there a correlation between myocardial deformation parameters of the left heart chambers with other important ultrasound parameters (eg maximal wall thickness, presence of subaortic obstruction, etc.) in patients with hypertrophic cardiomyopathy?
2. Is there a correlation between myocardial deformation parameters of the left heart chambers and the symptomatology or functional capacity of patients with hypertrophic cardiomyopathy?
3. Is there a correlation between the myocardial deformation parameters of the left heart chambers and the exercise capacity, as evidenced by the cardiopulmonary exercise test, in patients with hypertrophic cardiomyopathy?
4. Is there a correlation between myocardial deformation parameters of the left heart chambers with the risk of ventricular or supraventricular arrhythmias in patients with hypertrophic cardiomyopathy?
5. Is there a correlation between myocardial deformation parameters of the left heart chambers and risk factors for sudden death?

DETAILED DESCRIPTION:
Myocardial deformation parameters of the left heart chambers are of particular clinical importance because of their possible association with the severity of HCM and the presence of arrhythmias. However,current literature appears conflicting.

This is a prospective cohort study aiming to examine the echocardiographic parameters of myocardial deformation, estimated by the "speckle tracking" method, and their correlation with clinical presentation and symptomatology, other imaging parameters, exercise capacity, arrhythmias (ventricular or supraventricular) and risk factors for sudden death in patients with hypertrophic cardiomyopathy.

Although, similar efforts have been made in international literature, they are scarce and their results contradictory. The present study is the first to be performed in a Greek population, a fact that is particularly important given the genetic heterogeneity of the disease.

ELIGIBILITY:
Inclusion Criteria:

-Patients with diagnosed hypertrophic cardiomyopathy

Exclusion Criteria:

* Concomitant severe valvular heart disease
* Prior myocardial infarction
* History of atrial fibrillation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients with diagnosed hypertrophic cardiomyopathy that will proceed for assessment in AHEPA University Hospital. Only patients with severe valvular heart disease or prior myocardial infarction will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Cardiac arrest | 3 years
  Documented ventricular fibrillation or sustained ventricular tachycardia
Implantable cardioverter defibrillator therapy | 3 years
  Aproppriate Implantable cardioverter defibrillator therapy
All cause mortality | 3 years
  Death by any cause
Cardiovascular mortality | 3 years
  Death directly attributed to the primary disease

SECONDARY OUTCOMES:
Atrial fibrillation | 3 years
  Documented atrial fibrillation in patients with prior sinus rythm

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zegkos T, Parcharidou D, Ntelios D, Efthimiadis G, Karvounis H. The Prognostic Implications of Two-Dimensional Speckle Tracking Echocardiography in Hypertrophic Cardiomyopathy: Current and Future Perspectives. Cardiol Rev. 2018 May/Jun;26(3):130-136. doi: 10.1097/CRD.0000000000000172. PMID 29045290
- [Derived] Zegkos T, Ntelios D, Parcharidou D, Katranas S, Panagiotidis T, Papanastasiou CA, Karagiannidis E, Rouskas P, Vassilikos V, Karvounis H, Efthimiadis GK. The predictive value of left ventricular and left atrial mechanics for atrial fibrillation and heart failure in hypertrophic cardiomyopathy: a prospective cohort study. Int J Cardiovasc Imaging. 2021 Sep;37(9):2679-2690. doi: 10.1007/s10554-021-02232-0. Epub 2021 Apr 5. PMID 33818698